CLINICAL TRIAL: NCT00445848
Title: A Phase II Trial of the Combination of OSI-774 (Erlotinib; NSC-718781) and Bevacizumab (RHUMAB VEGF; NSC 704865) in Never-Smokers With Stage IIIB and IV Primary NSCLC Adenocarcinomas
Brief Title: S0636: Erlotinib and Bevacizumab in Never-Smokers With Stage IIIB or Stage IV Primary Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000531056; S0636 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib and Bevacizumab (Experimental)
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Biological: bevacizumab
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab also may stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Giving erlotinib together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving erlotinib together with bevacizumab works in treating patients with stage IIIB or stage IV primary non-small cell lung cancer who have never smoked.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess overall survival of patients with stage IIIB or IV primary non-small cell lung adenocarcinoma who have never smoked and are treated with erlotinib hydrochloride and bevacizumab.

Secondary

* Assess progression-free survival of patients treated with this regimen.
* Assess the response rate (confirmed and unconfirmed, complete and partial) in a subset of patients with measurable disease treated with this regimen.
* Evaluate the frequency and severity of toxicities associated with this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride daily on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Adenocarcinoma

    * No component of squamous cell carcinoma present
  * Incompletely resected or unresectable disease
* Stage IIIB or IV disease as defined below:

  * Selected stage IIIB disease

    * T4 (cytologically confirmed malignant pleural effusion OR pleural tumor foci that are separate from direct pleural invasion by the primary tumor)
    * Any N
    * M0
  * Stage IV disease

    * Any T
    * Any N
    * M1 (distant metastases present)
    * Recurrent lung cancer in a separate lobe after resection or radiotherapy within the past 5 years OR multifocal lesions in > 1 lobe considered stage IV disease
* New lesions occurring ≥ 5 years after resection may be considered a separate primary cancer and are not allowed if this is the only focus of lung cancer
* Measurable and/or nonmeasurable disease by CT scan, positron emission tomography scan, or MRI

  * Disease must be present outside a previous radiotherapy field OR a new lesion must be inside the port
  * Measurable disease must be assessed within the past 28 days
  * Nonmeasurable disease must be assessed within the past 42 days
  * Pleural effusions, ascites, and laboratory parameters are not acceptable as the only evidence of disease
* Must be a lifelong nonsmoker (< 100 cigarettes in lifetime)
* Treated brain metastases allowed provided the patient is asymptomatic and do not require steroids

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN if bone metastases present)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* Urine protein:creatinine ratio ≤ 0.5 OR urine protein < 1,000 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Hypertension allowed if controlled on medication prior to study enrollment
* Must be willing to provide prior smoking history
* No immediate life-threatening complications from malignancies
* No prior major medical condition, psychological condition, or social situation that would preclude study treatment
* No hemoptysis ≥ ½ teaspoon within the past 28 days
* No clinical history of pulmonary or upper respiratory hemorrhage ≥ grade 2 within the past 6 months or grade 1 within the past 28 days
* No history of either thrombosis or hemorrhage, including hemorrhagic or thrombotic stroke, or other CNS bleeding
* No serious nonhealing wound, ulcer, or bone fracture
* No other prior malignancy except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * In situ cervical cancer
  * Any other cancer from which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 7 days since prior fine-needle aspiration or core biopsy
* At least 28 days since prior radiotherapy (14 days for palliative radiotherapy) and recovered
* At least 28 days since prior surgery (e.g., thoracic or other major surgeries) and recovered
* At least 28 days since prior systemic chemotherapy
* Prior biologic therapy allowed
* No prior gefitinib, erlotinib hydrochloride, bevacizumab, or other targeted therapies against the epidermal growth factor receptor or vascular endothelial growth factor axes
* Concurrent stable, therapeutic anticoagulation therapy allowed (e.g., warfarin or low molecular weight heparin), provided the patient has no history of bleeding complications on anticoagulation or an inability to establish a stable therapeutic regimen for anticoagulation
* No concurrent surgery
* No other concurrent nonprotocol treatment (including chemotherapy, hormonal therapy, biological therapy, or radiotherapy) directed at this cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-07; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard L. West, MD, Study Chair — Swedish Cancer Institute at Swedish Medical Center - First Hill Campus
Locations (153):
- United States (153):
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Sutter Health - Western Division Cancer Research Group, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Central Dupage Cancer Center, Winfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Highland Hospital of Rochester, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Background] West HJ, Moon J, Hirsch FR, et al.: SWOG S0635 and S0636: Phase II trials in advanced-stage NSCLC of erlotinib (OSI-774) and bevacizumab in bronchioloalveolar carcinoma (BAC) and adenocarcinoma with BAC features (adenoBAC), and in never-smokers with primary NSCLC adenocarcinoma (adenoCa). [Abstract] J Clin Oncol 30 (Suppl 15): A-7517, 2012.
- [Result] Mack PC, Moon J, West HJ, et al.: Molecular marker analysis of SWOG S0636, a phase II trial of erlotinib and bevacizumab in never-smokers with advanced NSCLC. [Abstract] J Clin Oncol 30 (Suppl 15): A-7552, 2012.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 89 patients were enrolled. Four patients were excluded from the analysis: two patients were ineligible due to incorrect histology; two were no analyzable due to their not receiving any treatment on protocol.
Groups:
- Erlotinib and Bevacizumab: Patients received erlotinib 150 mg daily with bevacizumab at 15mg/kg until progression or prohibitive toxicity.
Period: Overall Study
Arm/Group | Erlotinib and Bevacizumab
Started | 85
Completed | 0
Not Completed | 85
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 4
Not completed — Progression | 62
Not completed — Other-Not protocol specified | 5

BASELINE CHARACTERISTICS:
Population: 85 patients were eligible and analyzable.
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 85
Age, Continuous [Median (Full Range); unit: years] | 61 [31 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 56
  African American | 4
  Asian | 21
  Native American | 2
  Unknown | 2
Performance Status [Number; unit: participants] — Patients with a SouthWest Oncology Group (SWOG) performance status (PS) of 0, 1, or 2 were eligible. Per protocol, PS = 0 Fully active, able to carry on all pre-disease performance without restriction; PS =1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work; PS = 2 Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  participants
    0/1 | 82
    2 | 3
Stage [Number; unit: participants] — Patients were required to have histologically proven stage IIIB (by pleural effusion) or IV lung adenocarcinoma as outlined below (AJCC Cancer Staging Manual, 6th Edition, 2002) Stage IIIB: T4, Any N, M0; Stage IV: Any T, Any N, M1. Any disease that is recurrent after surgery or radiation is classified as Stage IV.
  Following are more details about staging criteria:
  Any T: presence of tumor; T4: extensive tumor growth; Any N: lymph involvement; M0: no metastasis; M1: metastasis.
  participants
    IIIB(pleural effusion) | 15
    IV | 70

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Disease assessment is performed every 6 weeks for 18 weeks, then every 9-12 weeks until progression up to 2 years. After disease progression, patients must be followed every 3 months for 1 year and then every 6 months for a maximum of 3 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 85
months | 29.8 [22.5 to 37.8]
Statistical Analysis 1: Comparison: Erlotinib and Bevacizumab; The overall survival rate at year 1 was estimated using Kaplan-Meier; Test type: Other; proportion of participants = 0.78, 95% CI 2-sided [0.67 to 0.85]
Statistical Analysis 2: Comparison: Erlotinib and Bevacizumab; The overall survival rate at year 2 was estimated using Kaplan-Meier; Test type: Other; proportion of participants = 0.57, 95% CI 2-sided [0.46 to 0.67]
Statistical Analysis 3: Comparison: Erlotinib and Bevacizumab; The overall survival rate at year 3 was estimated using Kaplan-Meier; Test type: Other; proportion of participants = 0.43, 95% CI 2-sided [0.32 to 0.53]

2. Secondary Outcome: Progression-free Survival
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v 1.0), as a 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, or unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided) or appearance of any new lesion/site, or death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 85
months | 7.4 [6.1 to 10.9]

3. Secondary Outcome: Response Rate (Complete and Partial)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0): Complete Response (CR), Disappearance of all measurable and non-measurable disease; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: as for outcome 1
Population: Only patients with measurable disease at baseline were included in the analysis. 66 of 85 patients (78%) had measurable disease at baseline.
Measure: Number; unit: participants
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 66
participants
  Complete Response (CR) | 2
  Partial Response (PR) | 31
  Objective Response Rate (CR + PR) | 33
  Stable Disease (SD) | 23
  Non-Progression (ORR+SD) | 56
  Progressive Disease (PD) | 8
  Not Determinable/ Inadequate Assessment | 2

4. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 3.0. Only adverse events that are possibly, probably or definitely related to study drug are reported. Any CTCAE 3.0 event of Grade 3 (serious), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Time Frame: Toxicity assessment was evaluated after each cycle (21 days) while on protocol therapy.
Population: Eligible patients who had received the protocol treatments were included in the adverse event summaries.
Measure: Number; unit: Participants
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 85
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 3
  AST, SGOT | 4
  Anorexia | 1
  Bilirubin (hyperbilirubinemia) | 1
  Calcium, serum-low (hypocalcemia) | 1
  Colitis, infectious (e.g., Clostridium difficile) | 1
  Confusion | 2
  Dehydration | 1
  Dermatology/Skin-Other (Specify) | 1
  Diarrhea | 4
  Esophagitis | 1
  Fatigue (asthenia, lethargy, malaise) | 5
  Hemoglobin | 1
  Hemorrhage, GI - Stomach | 2
  Hemorrhage, pulmonary/upper respiratory - Lung | 1
  Hemorrhage, pulmonary/upper respiratory - Nose | 1
  Hypertension | 15
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 1
  Nail changes | 1
  Nausea | 2
  Neuropathy: motor | 1
  Pain - Abdomen NOS | 1
  Pain - Bone | 1
  Pain - Face | 1
  Pain - Joint | 1
  Potassium, serum-low (hypokalemia) | 1
  Proteinuria | 6
  Pruritus/itching | 1
  Rash/desquamation | 5
  Rash: acne/acneiform | 4
  Sodium, serum-low (hyponatremia) | 4
  Syncope (fainting) | 1
  Ulceration | 1
  Voice changes/dysarthria | 1
  Weight loss | 3

ADVERSE EVENTS:
Time Frame: Toxicity assessment was evaluated after each cycle (21 days) while on protocol therapy.
Arm/Group | Erlotinib and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 17/85
Other Adverse Events (participants affected / at risk) | 83/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Bevacizumab (N=85)
Hemoglobin (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1
Extremity-lower (gait/walking) (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Pain-Other (General disorders) | 1
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 3
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 3
Infection-Other (Infections and infestations) | 1
INR (of prothrombin time) (Investigations) | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Neuropathy: motor (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Bevacizumab (N=85)
Hemoglobin (Blood and lymphatic system disorders) | 19
Dry eye syndrome (Eye disorders) | 9
Ocular/Visual-Other (Eye disorders) | 6
Watery eye (epiphora, tearing) (Eye disorders) | 6
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 62
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 14
Flatulence (Gastrointestinal disorders) | 6
Heartburn/dyspepsia (Gastrointestinal disorders) | 13
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 7
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 8
Hemorrhoids (Gastrointestinal disorders) | 6
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 26
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 42
Pain - Abdomen NOS (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 20
Edema: limb (General disorders) | 14
Fatigue (asthenia, lethargy, malaise) (General disorders) | 55
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 7
Pain - Chest/thorax NOS (General disorders) | 12
Pain-Other (General disorders) | 12
Rigors/chills (General disorders) | 9
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 5
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 5
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 8
Infection-Other (Infections and infestations) | 9
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 25
AST, SGOT (Investigations) | 29
Alkaline phosphatase (Investigations) | 15
Bilirubin (hyperbilirubinemia) (Investigations) | 17
Creatinine (Investigations) | 20
Leukocytes (total WBC) (Investigations) | 11
Lymphopenia (Investigations) | 11
Metabolic/Laboratory-Other (Investigations) | 6
Weight loss (Investigations) | 28
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 26
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 5
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 5
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 24
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 10
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 16
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 7
Pain - Back (Musculoskeletal and connective tissue disorders) | 17
Pain - Bone (Musculoskeletal and connective tissue disorders) | 10
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 11
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 14
Pain - Joint (Musculoskeletal and connective tissue disorders) | 24
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 20
Pain - Neck (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 16
Neuropathy: sensory (Nervous system disorders) | 15
Ocular/Visual-Other (Nervous system disorders) | 6
Pain - Head/headache (Nervous system disorders) | 30
Taste alteration (dysgeusia) (Nervous system disorders) | 24
Insomnia (Psychiatric disorders) | 18
Mood alteration - anxiety (Psychiatric disorders) | 9
Mood alteration - depression (Psychiatric disorders) | 9
Glomerular filtration rate (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 21
Urinary frequency/urgency (Renal and urinary disorders) | 6
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 44
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 29
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 35
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 6
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 26
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 27
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 26
Nail changes (Skin and subcutaneous tissue disorders) | 12
Pruritus/itching (Skin and subcutaneous tissue disorders) | 23
Rash/desquamation (Skin and subcutaneous tissue disorders) | 43
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 63
Hemorrhage/Bleeding-Other (Vascular disorders) | 5
Hypertension (Vascular disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less